CLINICAL TRIAL: NCT00567853
Title: Clinical Investigation Of The Sorin 3D Annuloplasty Ring For Mitral Repair
Brief Title: Safety and Efficacy Study of the Sorin 3D Annuloplasty Ring For Mitral Repair
Acronym: MEMO3D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEMO3D.Reg
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Mitral Valve Regurgitation
Keywords: mitral valve regurgitation; mitral valve disease; mitral valve repair; mitral valve dysfunction; heart valve; valve disease; cardiac surgery
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEMO 3D ring (Other): All patients in the study will be implanted with the MEMO 3D ring
  Interventions: Device: Implantation of the MEMO 3D Annuloplasty Ring

INTERVENTIONS:
Device: Implantation of the MEMO 3D Annuloplasty Ring — Implantation of the MEMO 3D Annulopalsty Ring for mitral valve repair.

SUMMARY:
The purpose of this study is to collect data on the effectiveness and clinical outcomes of the MEMO 3D Annuloplasty ring as used for mitral valve repair.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years old or older
* An annuloplasty ring is indicated for reinforcement of a dysfunctional or diseased native mitral valve according to the current medical practice for valvular repair at each site.
* The subject is able to return for all follow-up evaluations of the study.

Exclusion Criteria:

* The subject or subject's legal representative is unwilling to sign the informed consent.
* The subject is or will be participating in another medical device or drug clinical trial.
* The subject is a minor, prisoner, institutionalized, or is unable to give informed consent.
* The subject has a life expectance of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with successful repair at 6 months. | One Year

SECONDARY OUTCOMES:
Freedom from re-operation at 12 months. Preoperative and postoperative mitral valve regurgitation and LV dimensions and mass assessed by echocardiography. Actuarial survival and freedom from clinical events at 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clark Hargrove, M.D., Principal Investigator — University of Pennsylvania Presbyterian Medical Center
Locations (6):
- United States (4):
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Pennsylvania Presbyterian Hospital, Philadelphia, Pennsylvania
  - The Heart Hospital Baylor Plano, Plano, Texas
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia